CLINICAL TRIAL: NCT02971215
Title: Effectiveness of High Intensity Laser Therapy in the Treatment of Subacromial Impingement Syndrome
Brief Title: Subacromial Impingement Syndrome Approach Using High Intensity Laser Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Castilla-La Mancha Health Service (Other); Hospital General Nuestra Señora del Prado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: jagHNSP
Record Dates: First submitted 2016-11-15; First posted 2016-11-22 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-03

CONDITIONS: Subacromial Impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-intensity laser therapy (Experimental): High-intensity laser therapy application through iLux Laser device
  Interventions: Device: iLux Laser
- Sham device (Sham Comparator): Sham high-intensity laser therapy application through sham iLux Laser device
  Interventions: Device: Sham ilux Laser

INTERVENTIONS:
Device: iLux Laser — Treatment during 15 sessions. It is divided in two phases: 1. 12W. 50 Hz 20% duty cycle. 50 J/cm² in painful zone. 2. 15 W. Burst (10 pulses-900 msec each train) 250 J/cm² in painful zone. Trough the iLux Laser (Mectronic Medicale, Italy)
  + Physical Therapy protocol.
  Arms: High-intensity laser therapy
Device: Sham ilux Laser — Sham treatment during 15 sessions trough the iLux Laser (Mectronic Medicale, Italy), It is applies the same time than experimental one but with 0 W + Physical Therapy protocol.
  Arms: Sham device

SUMMARY:
The purpose of this study is to assess the effectiveness of high intensity laser therapy in the treatment of subacromial impingement syndrome.

DETAILED DESCRIPTION:
Shoulder pain has a high prevalence in our society, several studies estimate an annual prevalence between 5% and 47%. It is one of the main causes of musculoskeletal pain, particularly in third place, after the low back pain and neck pain.

Symptoms of pathologies of subacromial space impingement syndrome, where, regardless of origin, pain is the number one symptom for the patient, which emanates functional impairment and the impact on quality of life. Because of the need to implement research to assess the effectiveness of high intensity laser therapy with new studies mayor methodological quality of obtaining conclusive results, and based on the scientific evidence supporting the low-power laser therapy as a useful tool in addressing the shoulder tendon pathology, we consider very interesting the realization of this research project.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 75 years old with diagnosis of subacromial impingement syndrome or any of the pathologies that compose it (tendinosis-tendinitis supraspinatus and rest of the rotator cuff, subacromial bursitis and tendinitis of the long head of the biceps).
* Visual Analogue Scale (VAS) less than or equal to 7.
* Forward flexion at least of 100º

Exclusion Criteria:

* Calcific tendinitis
* Complete rupture of the rotator cuff.
* Adhesive capsulitis.
* Clinical history of pathologies that without affecting the shoulder joint refer to painful shoulder symptoms (cervical root involvement, cervical surgery, cervical osteoarthritis and neurological pathologies)
* Fibromyalgia
* Be receiving physiotherapeutic treatment or have received it previously for this pathology one month before the start of treatment.
* Patients with alterations of thermal sensitivity.
* Derived from the absolute and relative contraindications of Laser Therapy:
* Photosensitive patients
* Neoplastic processes
* Hyperthyroidism
* Pregnancy
* Patients with a history of epileptic seizures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-11; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | Baseline
  SPADI test
Shoulder Pain and Disability Index (SPADI) | At the end of the laser protocol treatment (1 daily session during 15 workday -from monday to friday-)
  SPADI test
Shoulder Pain and Disability Index (SPADI) | one month after the end of the protocol treatment
  SPADI test
Shoulder Pain and Disability Index (SPADI) | three months after the end of the protocol treatment
  SPADI test
Constant-Murley Score | Baseline
  Constant-Murley Score without strength section. The results will be expressed on a maximum of 75 points.
Constant-Murley Score | At the end of the laser protocol treatment (1 daily session during 15 workday -from monday to friday-)
  Constant-Murley Score without strength section. The results will be expressed on a maximum of 75 points.
Constant-Murley Score | one month after the end of the protocol treatment
  Constant-Murley Score without strength section. The results will be expressed on a maximum of 75 points.
Constant-Murley Score | three months after the end of the protocol treatment
  Constant-Murley Score without strength section. The results will be expressed on a maximum of 75 points.
Quick-Dash Abbreviated | Baseline
  Quick- Dash Abbreviated test
Quick-Dash Abbreviated | At the end of the laser protocol treatment (1 daily session during 15 workday -from monday to friday-)
  Quick- Dash Abbreviated test
Quick-Dash Abbreviated | one month after the end of the protocol treatment
  Quick- Dash Abbreviated test
Quick-Dash Abbreviated | three months after the end of the protocol treatment
  Quick- Dash Abbreviated test

SECONDARY OUTCOMES:
Painful pressure threshold | Baseline, at the of the 15 sessions, one month after the end of the protocol treatment, three months after the end of the protocol treatment
  The pressure pain threshold will be measured by a pressure algometer and will be expressed in Newton.
Painful pressure threshold after first session | First session - 15 minutes after laser or sham treatment.
  The pressure pain threshold will be measured by a pressure algometer and will be expressed in Newton.
VAS | Baseline, at the of the 15 sessions, one month after the end of the protocol treatment, three months after the end of the protocol treatment
  Visual analogue scale

OTHER OUTCOMES:
Quality of life | Baseline
  EQ-5D™ is a standardised instrument for use as a measure of health outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Aceituno-Gomez, PT, Principal Investigator — Castilla-La Mancha Health Service
Locations (1):
- Hospital General Nuestra Señora del Prado, Talavera de la Reina, Toledo, Spain